CLINICAL TRIAL: NCT01425151
Title: The i-GelTM. A Randomized, Crossover Study With the Laryngeal Mask Airway ProSealTM in Anesthetized Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, ChristianKeller, MD, M.Sc., Schulthess Klinik
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Schulthess_Anä_2
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Device Success Rate; Device Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- i-Gel (Active Comparator)
  Interventions: Device: i-Gel
- ProSeal (Experimental)
  Interventions: Device: ProSeal

INTERVENTIONS:
Device: i-Gel — Oropharyngeal leak pressure Insertion success
  Arms: i-Gel
Device: ProSeal — Oropharyngeal leak pressure Insertion success
  Arms: ProSeal

SUMMARY:
In the following randomized, crossover study, the investigators test the hypothesis that ease of insertion and oropharyngeal leak pressure differ between the LMA ProSealTM and the i-GelTM in anesthetized pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Age 1.5-6 years

Exclusion Criteria:

* known or predicted difficult airway
* body mass index > 35 kg m-2
* risk of aspiration

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 10 Minutes

SECONDARY OUTCOMES:
Insertion success rate | 1 Minute

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD, M.Sc., Principal Investigator — Schulthess Klinik
Locations (2):
- Klinik für Anästhesie und Allgemeine Intensivmedizin, Innsbruck, Austria
- Christian Keller, Zurich, Switzerland